CLINICAL TRIAL: NCT06304675
Title: Manageable Environmental Factors Affect Treatment Response as Much as Migraine Phenotype
Brief Title: Manageable Environmental Factors in Migraine
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Bilge Piri Cinar, Professor of Clinic, Samsun University
Other Study IDs: 905055423985
Record Dates: First submitted 2024-02-06; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
There is limited and insufficient information on the effects of inappropriate living environments, exposure to allergens, electromagnetic fields and stress factors on the chronicity of migraine. The aim of this study is to investigate the frequency of environmental variables/triggers in episodic and chronic migraine patients and their relationship with clinical variables in the chronic migraine group. The results obtained will be shared not only in the scientific community, but also on workplace health and employer-related platforms, including "Wellbeing" groups.

DETAILED DESCRIPTION:
Migraines are a prevalent and debilitating neurological condition that can significantly impact a person's quality of life. While various genetic and environmental factors contribute to the development and progression of migraines, the role of specific environmental factors/triggers in the chronification of this condition remains inadequately explored. This paper seeks to address this research gap by focusing on the impact of inadequate living environments, exposure to allergens, electromagnetic fields, and stressors on the chronification of migraines.

Obtaining specific trigger and headache information from a large number of migraineurs may provide a better understanding of which triggers are common and/or strong and which may become important only when they act together (6). With studies focusing on this issue, data that will even enable the identification of individuals with migraine who share a set of common triggers can be obtained.

Migraine attacks often begin with an episodic course and may become chronic in some individuals over time due to reasons such as drug overuse, various environmental factors and failure to take necessary steps in lifestyle regulation. Exactly when chronicity will begin in each individual and how it will progress are related to these endogenous and exogenous factors as well as the genetic structure of the individual, and how it will progress cannot be predicted.

It is difficult to study the effect of triggers on migraine attacks. Possible triggers may interact and statistical modeling is often difficult. Therefore, the estimated frequencies of precipitating factors vary considerably depending on the study approach and population. There are very few studies investigating the effects of trigger and environmental factors on the migraine phenotype. In a study where episodic and chronic migraine groups and trigger/environmental factors were evaluated in 300 women with migraine; Although some triggers have been defined for migraine, no differentiation was observed between episodic and chronic migraine groups. However, in a study conducted in 2023, endogenous and exogenous factors that may have an effect on the chronicity of migraine were evaluated. Although some triggers/environmental factors have been identified as risk factors, their likelihood of co-occurrence and clustering have not been evaluated in a large population.

In this study, the effects of triggers and environmental factors, which investigators identified with a comprehensive inquiry form, on both the pain phenotype and treatment response in migraine cases followed up in the same clinic, including episodic and chronic migraine cases, were evaluated. It is aimed to show how these factors come together in the episodic and chronic migraine group and how this affects the fate of the patient as well as the fate of the pain. Additionally, the relationship between treatment options for migraine and the responses received and environmental factors/triggers was investigated. Researching and defining all these features may be a good predictor in the chronicity of migraine, which affects many individuals, and in the regulation of environmental factors/triggers.

Materials and Methods:

Participants: Patients who were over 18 years of age, were followed up with a diagnosis of migraine, and had the cognitive level to provide information about demographic and clinical features of headache were included. International Classification of Headache Disorders-3 (ICHD-3) criteria were used for the diagnosis of chronic migraine in the study group. Having a headache more than 15 days per month for >3 months and having at least 8 headaches with migraine characteristics was defined as "chronic migraine", while those with headaches less frequently than 14 days per month were defined as "episodic migraine". All treatment options and responses received for migraine were recorded in detail. Participants who agreed to participate in the study were given a survey form containing items about migraine characteristics, triggers and environmental factors. The data form was filled in through a face-to-face interview.

2.2. Study Design: Ethics approval was received for this cross-sectional-observational study (OndokuzMayısUniversity-OMU-2023/466). The International Headache Society (IHS) is involved in the development and publication of numerous guidelines for controlled treatment trials for primary headache disorders. In the planning and implementation stages of this study, the clinical trials guideline principles of the I IHS were followed and progress was made according to the STROBE checklist. The demographic characteristics of the patients were recorded in the demographic data form. Then, the patient's headache characteristics (duration, type, presence of aura, accompanying features, etc.) and the answers to questions about possible triggers of migraine and environmental factors were recorded in the data form.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between 18-70 years old
2. Clinical diagnosis of migraine
3. Cognitive level to provide information about demographic and clinical features of headache

Exclusion Criteria:

1) Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with migraine in the neurology clinic and followed up with this diagnosis and who agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
1. Environmental factors/triggers affecting the chronicity of migraine | 3-months
  Triggers/environmental factors in individuals diagnosed with chronic migraine and episodic migraine were documented with an inquiry-survey form and demographic data form.
  (The inquiry form/survey form containing the list of triggers/environmental factors can be uploaded to the system if desired) There is no scoring system in this inquiry form/survey form.

SECONDARY OUTCOMES:
2.Environmental factors/triggers and migraine treatment | 3-months
  Environmental factors/triggers that may affect migraine treatment success were evaluated with a survey form.
  (The inquiry form/survey form containing the list of triggers/environmental factors can be uploaded to the system if desired) There is no scoring system in this inquiry form/survey form.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data with a similar study plan can be shared within the scope of a study for big data or review/meta analysis

REFERENCES:
- [Result] Spierings EL, Donoghue S, Mian A, Wober C. Sufficiency and necessity in migraine: how do we figure out if triggers are absolute or partial and, if partial, additive or potentiating? Curr Pain Headache Rep. 2014 Oct;18(10):455. doi: 10.1007/s11916-014-0455-y. PMID 25163437
- [Result] Guidelines for controlled trials of drugs in migraine. First edition. International Headache Society Committee on Clinical Trials in Migraine. Cephalalgia. 1991 Feb;11(1):1-12. No abstract available. PMID 2036663
- [Result] Tfelt-Hansen P, Block G, Dahlof C, Diener HC, Ferrari MD, Goadsby PJ, Guidetti V, Jones B, Lipton RB, Massiou H, Meinert C, Sandrini G, Steiner T, Winter PB; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: second edition. Cephalalgia. 2000 Nov;20(9):765-86. doi: 10.1046/j.1468-2982.2000.00117.x. No abstract available. PMID 11167908
- [Result] Hajjarzadeh S, Shalilahmadi D, Nikniaz Z, Mahdavi R, Hajjarzadeh S. The comparison of the main dietary and non-dietary trigger factors in women with chronic and episodic migraine. Nutr Diet. 2022 Nov;79(5):616-622. doi: 10.1111/1747-0080.12761. Epub 2022 Aug 18. PMID 35983599
- [Result] Lipton RB, Buse DC, Nahas SJ, Tietjen GE, Martin VT, Lof E, Brevig T, Cady R, Diener HC. Risk factors for migraine disease progression: a narrative review for a patient-centered approach. J Neurol. 2023 Dec;270(12):5692-5710. doi: 10.1007/s00415-023-11880-2. Epub 2023 Aug 24. PMID 37615752